CLINICAL TRIAL: NCT06177782
Title: Accuracy of Tooth Modified Scan Bodies as a Novel Technique for Edentulous Full Arch Implant Supported Dental Prosthesis: A Controlled Clinical Trial
Brief Title: Accuracy of Tooth Modified Scan Bodies as a Novel Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Adel Salah Khattab, Associate Professor, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22859
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Digital Technology; Dental
Keywords: Jaw relation; Scan body

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tooth Modified Scan Bodies (Active Comparator): The intraoral scanner (IOS) impression will be recorded using modified scan bodies. The IOS device will be calibrated right before the impression. The scan strategy will be consistent for all the procedures following the manufacturer guidelines.
  Interventions: Device: Tooth modified scan bodies
- Conventional Scan Bodies (Placebo Comparator): The intraoral scanner (IOS) impression will be recorded using conventional implant scan bodies secured at the multiunit abutment level.
  Interventions: Device: Conventional scan bodies

INTERVENTIONS:
Device: Tooth modified scan bodies — Tooth modified scan bodies are used during scanning for full arch implant cases.
  Arms: Tooth Modified Scan Bodies
Device: Conventional scan bodies — Conventional scan bodies will be used for scanning the full arch implant cases.
  Arms: Conventional Scan Bodies

SUMMARY:
The clinical performance of a novel scan body Tooth Modified Scan Body (TMSB) in the degree of trueness of IOS impression for full arch cases.

I

DETAILED DESCRIPTION:
The clinical performance of a novel scan body Tooth Modified Scan Body (TMSB) in the degree of trueness of IOS impression for full arch cases. TMSB is a scan body to which different teeth are attached directly as one piece, this may enhance the accuracy level by filling the gabs between ISB as well as acting as a stable artificial AI-easily recognized landmarks thus facilitating the scanning procedure. OS impression utilizing tooth modified scan bodies or conventional scan bodies result in the same degree of trueness as conventional verified splinted open tray impression. To our knowledge, it is the first time in the literature to utilize a novel scan body modified with directly connected teeth as artificial landmarks in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Participants who had received 4-6 implants in 1 edentulous arch.
* Participants with 1-piece implant-supported complete-arch fixed dental prostheses.
* Systemically free.
* Primary implant stability exceed 72 the day of the definitive impression.

Exclusion Criteria:

* Smoker's.
* Non co-operative patients.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Degree of trueness | Immediately postoperative
  Digital files will be obtained: either conventional scan or TMSB scan. All the STL files will be imported to dental CAD software , and scan bodies will be converted to implant multi-unit ti-base replicas using a digital library. Then, updated STL files will be imported to inspection software for trueness assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

REFERENCES:
- [Derived] Eldabe AK, Adel-Khattab D, Botros KH. Trueness of tooth modified scan bodies as a novel technique for edentulous full arch implant supported dental prosthesis: an in vivo prospective comparative study. BMC Oral Health. 2025 Jan 6;25(1):29. doi: 10.1186/s12903-024-05172-y. PMID 39762850